CLINICAL TRIAL: NCT01490996
Title: A Phase I/IIa Study Combining Curcumin (Curcumin C3-Complex, Sabinsa) With Standard Care FOLFOX Chemotherapy in Patients With Inoperable Colorectal Cancer.
Brief Title: Combining Curcumin With FOLFOX Chemotherapy in Patients With Inoperable Colorectal Cancer
Acronym: CUFOX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0225
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2017-05

CONDITIONS: Colonic Cancer; Metastasis
Keywords: Curcumin; Colorectal cancer; metastases; FOLFOX
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis; Colorectal Neoplasms | interventions — Drug Therapy; Curcumin; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy only (Active Comparator): Patients receiving up to 12 cycles of therapy. Standard care pathway management.
  Interventions: Drug: Chemotherapy only
- Chemotherapy plus curcumin (Experimental): Patients taking daily oral curcumin for up to 12 cycles of therapy. Standard care pathway management.
  Interventions: Drug: Oral complex C3 curcumin + chemotherapy

INTERVENTIONS:
Drug: Oral complex C3 curcumin + chemotherapy — Daily oral capsule(s)
  Other Names: C3-complex curcumin (diferuloylmethane)
  Arms: Chemotherapy plus curcumin
Drug: Chemotherapy only — Standard care chemotherapy
  Other Names: FOLFOX (protocol includes changes to XELOX - capecitabine)
  Arms: Chemotherapy only

SUMMARY:
Oral curcumin (complex C3, Sabinsa Corp, Utah) will be given to patients with inoperable colorectal metastases who will be commencing standard care oxaliplatin-based (FOLFOX) chemotherapy for up to 12 cycles(approximately 6 months) of treatment.

Primary measurements focus on safety and tolerability. These will be recorded in real-time and report the number and severity of adverse events.

Secondary measurements will include efficacy, (measured by response rate with RECIST and overall survival in months) supported by biomarker analysis.

DETAILED DESCRIPTION:
Hypothesis Combination of oral curcumin with FOLFOX-based chemotherapy will be a safe and tolerated regimen for long-term administration to patients with colorectal metastases.

Primary objectives

To establish a tolerated dose of daily oral curcumin to be taken long-term with FOLFOX-based chemotherapy in patients with metastatic colorectal cancer will be conducted to assess:

1. Safety, tolerability and feasibility of administering oral curcumin at increasing doses escalating to 4 capsules (≈2 g C3-complex) during FOLFOX-based chemotherapy and continued for the duration of the chemotherapy course.

Secondary objectives

1. To observe any changes to the neuropathic side-effects of chemotherapy.
2. To observe potential for efficacy in terms of disease response and survival.
3. To identify putative biomarkers in plasma.

This is a phase I/IIa study:

Phase I will be a traditional escalation response design study (or 3+3+3) to firstly assess the safety of this combination and identify a maximum tolerated dose up to 4 g per day.

Phase IIa will be a randomised control study comparing curcumin and FOLFOX with FOLFOX alone, recruited at a 2:1 ratio respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of metastatic colorectal cancer
* Measurable disease by Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) (Appendix 1)
* Adequate haematological, hepatic and renal function
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1
* Patients must have recovered from effects of any recent major surgery
* Willing to use contraception if applicable
* Informed consent
* Life expectancy estimated to be more than 12 weeks

Exclusion Criteria:

* Main exclusion criteria
* Contraindications to FOLFOX chemotherapy: Peripheral neuropathy NCI CTC >1, Liver failure, uncontrolled coronary heart disease, myocardial infarction within the previous 6 months.
* Unwilling or unable to comply with the study protocol.
* Patients who are pregnant or lactating or contemplating pregnancy. Patients or their partners who become pregnant during the study will be referred to the appropriate experts.
* Undergone chemotherapy (other than adjuvant for CRC) or participating in another drug study.
* Previous cancer <5 years (other than colorectal, basal cell carcinoma, in-situ cervical cancer).
* Major surgery within 4 weeks of starting the study
* Co-existing active infection or serious concurrent medical condition
* Significant cardiovascular disease
* Bone metastases
* Known brain or leptomeningeal metastases
* Surgery or hospital admissions for symptomatic intra-abdominal adhesions
* Active endoscopically proven peptic ulcer disease or colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-02; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Completion of dose escalation over 2 cycles of therapy | 1 year
  Patients will start curcumin a week prior to chemotherapy. Upon completion of two cycles of therapy without dose-limiting toxicity in 3 consecutive patients, the dose will be escalated for the next 3 patients. Real-time adverse event reporting will be undertaken to record number and severity of events.

SECONDARY OUTCOMES:
Completion of (or withdrawal from) chemotherapy | Up to 6 months
  Compliance in the study will be measured in months/cycles of therapy tolerated. Reasons for withdrawal or cessation will be documented which will include mortality, adverse events and patient reported outcomes of tolerance to the protocol regimen.
Efficacy in terms of disease response and survival | Up to 7 years
  Response rate will be measured using RECIST. Overall survival will be measured in months.

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Thomas, PhD FRCS, Principal Investigator — University of Leicester/University Hospitals Leicester
Locations (1):
- Dept Oncology, Leicester Royal Infirmary, Leicester, United Kingdom

REFERENCES:
- [Derived] Howells LM, Iwuji COO, Irving GRB, Barber S, Walter H, Sidat Z, Griffin-Teall N, Singh R, Foreman N, Patel SR, Morgan B, Steward WP, Gescher A, Thomas AL, Brown K. Curcumin Combined with FOLFOX Chemotherapy Is Safe and Tolerable in Patients with Metastatic Colorectal Cancer in a Randomized Phase IIa Trial. J Nutr. 2019 Jul 1;149(7):1133-1139. doi: 10.1093/jn/nxz029. PMID 31132111
- [Derived] James MI, Iwuji C, Irving G, Karmokar A, Higgins JA, Griffin-Teal N, Thomas A, Greaves P, Cai H, Patel SR, Morgan B, Dennison A, Metcalfe M, Garcea G, Lloyd DM, Berry DP, Steward WP, Howells LM, Brown K. Curcumin inhibits cancer stem cell phenotypes in ex vivo models of colorectal liver metastases, and is clinically safe and tolerable in combination with FOLFOX chemotherapy. Cancer Lett. 2015 Aug 10;364(2):135-41. doi: 10.1016/j.canlet.2015.05.005. Epub 2015 May 12. PMID 25979230
- [Derived] Irving GR, Iwuji CO, Morgan B, Berry DP, Steward WP, Thomas A, Brown K, Howells LM. Combining curcumin (C3-complex, Sabinsa) with standard care FOLFOX chemotherapy in patients with inoperable colorectal cancer (CUFOX): study protocol for a randomised control trial. Trials. 2015 Mar 24;16:110. doi: 10.1186/s13063-015-0641-1. PMID 25872567